CLINICAL TRIAL: NCT02754245
Title: A Validation Study of Emergency Department Crowding Estimation
Brief Title: ED Overcrowding Validation Study
Acronym: EDOVS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Collaborators: JPS Health Network (Other); Baylor University (Other)
Responsible Party: Sponsor
Other Study IDs: 014-013
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Emergency Department Overcrowding
Keywords: multicenter study; emergency department; overcrowding status; estimation tool; validation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- JPS: study sample at JPS included for analysis
- BUMC Dallas: study sample at Baylor University Medical Center Dallas included for analysis
- BUMC at Gardin: study sample at Baylor University Medical Center Gardin included for analysis
- BUMC Waxahachie: study sample at Baylor University Medical Center Waxahachie included for analysis
- BUMC Carrolton: study sample at Baylor University Medical Center Carrolton included for analysis
- BUMC McKinney: study sample at Baylor University Medical Center McKinney included for analysis

SUMMARY:
The aim of this study is to externally validate a new emergency department overcrowding estimation tool (SONET) developed at John Peter Smith Health Network (JPS).

DETAILED DESCRIPTION:
In recent years, emergency department (ED) overcrowding has become more and more common in regional and tertiary referral hospitals. ED overcrowding status significantly affects ED operational efficiency, resulting in ambulance diversion, increased ED 72h return visits, patient satisfaction, and left without being seen (LWBS) rates.

Several estimation tools were derived to determine ED overcrowding status using various operational parameters such as, but not limited to, total number of ED patients, total ED admission holds, nursing staff, and patient injury severity. However, these tools cannot precisely evaluate ED overcrowding status, nor show strong correlations with ED operational inefficiency. The National Emergency Department Overcrowding Study (NEDOCS) is a widely used estimation tool to determine ED overcrowding status with relatively high consistency rates. However, the study was not able to evaluate interrater reliability since no standard definition of overcrowding existed.

An ED overcrowding estimation tool, SONET, was developed and internally validated at JPS and showed more consistency and accuracy when compared to estimation rates utilizing NEDOCS. All things considered, it is worthwhile to perform a survey study to determine the interrater variability between different evaluators for an ED overcrowding evaluation tool, one utilizing all possible collectible operational variables. In order to minimize the bias and further determine the accuracy of evaluating ED overcrowding status, a multi-center external validation study is warranted. This study will extend to six sites for the purpose of externally validating JPS' novel ED overcrowding estimation tool, SONET, by comparing its overcrowding estimation rates with those derived utilizing NEDOCS.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients visiting the emergency department or urgent care clinic at any one of the six participating sites during the allocated one month time period

Exclusion Criteria:

* those who do not meet inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients visiting any one of the six participating sites (one JPS ED or urgent care clinic or one of five Baylor emergency departments or urgent care clinics) during the allocated one month time period
Sampling Method: Probability Sample
Enrollment: 55000 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
left without being seen disposition chart review | 30 days
  LWBS refers to patients who have been called at least three times, using 20 minute intervals, to occupy an ED exam bed, however, do not respond. If after the third attempt the patient responds, the investigators will consider this a new patient registration/encounter. These data will be collected for each patient during the study period during initial ED registration and upon ED disposition.
emergency department 72 hour return chart review | 30 days
  ED 72h return will be defined to patients who re-register to the same ED as a new patient (unplanned) within 72h of a previous departure, regardless of the complaint. Planned ED revisits within 72h will be excluded. These data will be collected during initial ED registration during study period and will follow up each patient at least 72h post-discharge.
emergency department mortality | 30 days
hospital mortality | 30 days
emergency department length of stay | 30 days

SECONDARY OUTCOMES:
patient satisfaction survey | 30 days
  Patient satisfaction will be measured using Qualitick (Clearwater, FL), a real-time patient satisfaction program reporting tool using a Likert scale format. Patient will complete their Qualitick survey upon departure from ED regardless of their ED dispositions (e.g. transfer to inpatient service, discharge to home, transfer to another facility, etc.). Patients, or patient designees, will use a tablet to answer a series of questions. Patients, or their designees, have the option of omitting their name to ensure their information is kept anonymous.
physician empathy scale | 30 days
  Jefferson Physician Empathy Scale, available online, will be conducted by ED staff and compared with 1) staff working different shifts with different levels of crowding; 2) the norms; 3) staff working a more balanced schedule (roughly equal numbers of day, evening, and night shifts); and 4) attending physicians versus nursing staff versus residents. Average scores will be used to determine any differences among groups. The measurement tool will be repeated 6-9 months later to determine whether dynamic changes have occurred and whether an association exists with respect to changes in operation efficiency as a function of relative ED crowding at the individual physician level during the study period. The investigators recognize that the inclusion of the psychometric tests will be, to some extent, exploratory and the most important assessment will be the simple descriptive display of the mean scores (and standard deviations).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein SL, Verghese V, Leung W, Lunney AT, Perez I. Development and validation of a new index to measure emergency department crowding. Acad Emerg Med. 2003 Sep;10(9):938-42. doi: 10.1111/j.1553-2712.2003.tb00647.x. PMID 12957975
- [Background] Weiss SJ, Derlet R, Arndahl J, Ernst AA, Richards J, Fernandez-Frackelton M, Schwab R, Stair TO, Vicellio P, Levy D, Brautigan M, Johnson A, Nick TG. Estimating the degree of emergency department overcrowding in academic medical centers: results of the National ED Overcrowding Study (NEDOCS). Acad Emerg Med. 2004 Jan;11(1):38-50. doi: 10.1197/j.aem.2003.07.017. PMID 14709427
- [Background] Epstein SK, Tian L. Development of an emergency department work score to predict ambulance diversion. Acad Emerg Med. 2006 Apr;13(4):421-6. doi: 10.1197/j.aem.2005.11.081. PMID 16581932
- [Background] McCarthy ML, Aronsky D, Jones ID, Miner JR, Band RA, Baren JM, Desmond JS, Baumlin KM, Ding R, Shesser R. The emergency department occupancy rate: a simple measure of emergency department crowding? Ann Emerg Med. 2008 Jan;51(1):15-24, 24.e1-2. doi: 10.1016/j.annemergmed.2007.09.003. Epub 2007 Nov 5. PMID 17980458
- [Background] Jones SS, Allen TL, Flottemesch TJ, Welch SJ. An independent evaluation of four quantitative emergency department crowding scales. Acad Emerg Med. 2006 Nov;13(11):1204-11. doi: 10.1197/j.aem.2006.05.021. Epub 2006 Aug 10. PMID 16902050
- [Background] Wang H, Robinson RD, Garrett JS, Bunch K, Huggins CA, Watson K, Daniels J, Banks B, D'Etienne JP, Zenarosa NR. Use of the SONET Score to Evaluate High Volume Emergency Department Overcrowding: A Prospective Derivation and Validation Study. Emerg Med Int. 2015;2015:401757. doi: 10.1155/2015/401757. Epub 2015 Jun 8. PMID 26167302